CLINICAL TRIAL: NCT03464630
Title: Reducing Maternal Depression and Promoting Infant Social-Emotional Health & Development
Acronym: MBN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgia State University (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Oregon Research Institute (Other); The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kathleen Baggett, Associate Professor, Georgia State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01HD086894 (NIH); R01HD086894-01A1 (NIH)
Record Dates: First submitted 2018-02-28; First posted 2018-03-14 (Actual); Results first posted 2024-06-20 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-05

CONDITIONS: Maternal Depression and Parent Practices, Postpartum; Infant Development
Keywords: Treatment Maternal depression postpartum; Optimizing Maternal parenting practices; Optimizing Infant development; Optimizing Infant behavior; Direct observation of mother-Infant interaction; M health intervention; Remote coaching; RCT

STUDY DESIGN:
Intervention Model Description: Two arm, randomized controlled intent to treat trial
Who Masked: Participant, Outcomes Assessor
Masking Description: Assessment coders and participants are naive to treatment condition
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mom & Baby Net (Experimental): CBT skills based mobile intervention targeting maternal depression and sensitive responsive parenting practices for optimizing infant social-communication promotion and provision of community resources and referral
  Interventions: Behavioral: Mom & Baby Net
- Depression & Developmental Awareness System (Active Comparator): Supportive, person-centered mobile intervention targeting maternal awareness of maternal depression symptoms, infant developmental milestones, and provision of community resources and referral (active control condition)
  Interventions: Behavioral: Depression & Developmental Awareness System

INTERVENTIONS:
Behavioral: Mom & Baby Net — CBT skills based mobile intervention targeting maternal depression and sensitive responsive parenting practices for optimizing infant social-communication promotion and provision of community resources and referral
  Arms: Mom & Baby Net
Behavioral: Depression & Developmental Awareness System — Supportive, person-centered mobile intervention targeting maternal awareness of maternal depression symptoms, infant developmental milestones, and provision of community resources and referral (active control condition)
  Arms: Depression & Developmental Awareness System

SUMMARY:
A mobile remote coaching program study to improve maternal mood and increase parenting practices that lead to better infant social-emotional and communication outcomes

DETAILED DESCRIPTION:
To address the life course needs of depressed mothers and their infants, brief, accessible, and integrated interventions that target both maternal depression and specific nurturing parent behaviors demonstrated to improve infant social-emotional communication outcomes are needed. In prior programmatic research, two separate web-based, remote coaching interventions for: (a) parent nurturing behaviors that improve infant outcomes (Baby-Net R34; R01) [13], and (b) maternal depression (Mom-Net R34; R01) [14] were developed. Compared to controls, the Baby-Net program demonstrated medium to large effects on observed nurturing parent behavior and on infant social-emotional competencies in the context of play [13] and in the context of book activities [15]. Mom-Net demonstrated low attrition and high levels of feasibility, program use, and satisfaction [14]. Compared to controls, Mom-Net participants demonstrated significant reductions in depression and improved preschool parenting behavior [14]. A substantial advantage of the mobile, remote coaching approach is that it overcomes multiple logistical barriers that often prevent low-income mothers from participating in community/home visiting treatment programs [2]. Thus, this prior research on web-based maternal depression and specific nurturing parenting behavior in infancy, provides a strong empirical basis for the Mom & Baby Net program. Investigators will rigorously test the merged Mom & Baby Net intervention effects with a total sample of 368 participants (184 mothers with depression and 184 infants) via a 2-arm, intent-to-treat, randomized controlled trial.

The start date of this grant-funded randomized controlled trial was September 1, 2016. Data collection is currently underway and scheduled to conclude in March 2022. Following IRB-approved pilot work, the randomized controlled trial was IRB- approved on November 17, 2017. Immediately following IRB approval, recruitment was initiated. Between February 15, 2018 and March 11, 2021, we successfully consented a total sample of 368 participants (184 women and 184 infants) into the randomized controlled trial. The sample is predominantly Black and socioeconomically disadvantaged.

ELIGIBILITY:
Inclusion Criteria:

* Mother is 18 years of age
* Mother speaks English
* Mother lives in metro-Atlanta area
* Mother has baby younger than 12 months of age
* Mother has positive depression screen (PHQ2)

Exclusion Criteria:

Stressors that mother specifies at the time of screening that would interfere with study participation such as: maternal homelessness, mental or physical health condition (diagnosed with schizophrenia or treatment/medication for hallucinations/delusions), current inpatient treatment for mental health or substance abuse. Infant exclusion criteria include factors that could render research participation stressful, such as intensive treatment for a genetic or health condition or not in permanent legal guardian custody

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Baggett, PhD, Principal Investigator — Georgia State University
Locations (1):
- Georgia State University, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baggett KM, Davis B, Mosley EA, Miller K, Leve C, Feil EG. Depressed and Socioeconomically Disadvantaged Mothers' Progression Into a Randomized Controlled Mobile Mental Health and Parenting Intervention: A Descriptive Examination Prior to and During COVID-19. Front Psychol. 2021 Aug 12;12:719149. doi: 10.3389/fpsyg.2021.719149. eCollection 2021. PMID 34456828
- [Background] Baggett KM, Davis B, Sheeber LB, Ammerman RT, Mosley EA, Miller K, Feil EG. Minding the Gatekeepers: Referral and Recruitment of Postpartum Mothers with Depression into a Randomized Controlled Trial of a Mobile Internet Parenting Intervention to Improve Mood and Optimize Infant Social Communication Outcomes. Int J Environ Res Public Health. 2020 Dec 2;17(23):8978. doi: 10.3390/ijerph17238978. PMID 33276610
- [Background] Baggett KM, Davis B, Sheeber L, Miller K, Leve C, Mosley EA, Landry SH, Feil EG. Optimizing Social-Emotional-Communication Development in Infants of Mothers With Depression: Protocol for a Randomized Controlled Trial of a Mobile Intervention Targeting Depression and Responsive Parenting. JMIR Res Protoc. 2021 Aug 18;10(8):e31072. doi: 10.2196/31072. PMID 34406122

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participant flow shows 368 total participants enrolled, which matches the Protocol section documenting 368 total participants enrolled
Period: Overall Study
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Started (Consented, pre-assessed, & randomized) | 184 (92 mothers and 92 infants) | 184 (92 mothers and 92 infants)
Initiated & Completed Orientation Session | 172 (86 mothers and 86 infants) | 182 (91 mothers and 91 infants)
Initiated & Completed S1 Intervention Content | 170 (85 mothers and 85 infants) | 172 (86 mothers and 86 infants)
Initiated Post-Assessment | 142 (71 mothers and 71 infants) | 158 (79 mothers and 79 infants)
Completed (Initiated & completed 6-month Follow Up) | 98 (49 mothers and 49 infants) | 118 (59 mothers and 59 infants)
Not Completed | 86 | 66
Not completed — Lost to Follow-up | 62 | 52
Not completed — Withdrawal by Subject | 16 | 10
Not completed — Passive Disengagement | 8 | 4

BASELINE CHARACTERISTICS:
Population: Participant dyads (mothers and infants) who consented and completed pre-assessment
Groups:
- Total: Total of all reporting groups
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System | Total
Number analyzed (Participants) | 184 | 184 | 368
Age, Categorical [Count of Participants; unit: Participants] — Population: Age for one participant dyad is unknown
  Participants
    Mothers: number analyzed (Participants) | 91 | 92 | 183
    Mothers: <=18 years | 0 | 0 | 0
    Mothers: Between 18 and 65 years | 91 | 92 | 183
    Mothers: >=65 years | 0 | 0 | 0
    Infants: number analyzed (Participants) | 91 | 92 | 183
    Infants: <=18 years | 91 | 92 | 183
    Infants: Between 18 and 65 years | 0 | 0 | 0
    Infants: >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Age for one participant dyad is unknown. Mother and infant age are reported separately - infant age is reported in years and not months since we are unable to indicate two units of measure.
  years
    Mothers: number analyzed (Participants) | 91 | 92 | 183
    Mothers | 27.63 (5.90) | 28.58 (5.71) | 28.11 (5.81)
    Infants: number analyzed (Participants) | 91 | 92 | 183
    Infants | 0.51 (0.25) | 0.50 (0.23) | 0.50 (0.24)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One participant did not report their infant's gender
  Participants
    Mothers: number analyzed (Participants) | 91 | 92 | 183
    Mothers: Female | 91 | 92 | 183
    Mothers: Male | 0 | 0 | 0
    Infants: number analyzed (Participants) | 91 | 92 | 183
    Infants: Female | 44 | 48 | 92
    Infants: Male | 47 | 44 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Ethnicity for one mother/infant dyad was not reported
  Participants
    Mothers: number analyzed (Participants) | 92 | 92 | 184
    Mothers: Hispanic or Latino | 1 | 4 | 5
    Mothers: Not Hispanic or Latino | 90 | 88 | 178
    Mothers: Unknown or Not Reported | 1 | 0 | 1
    Infants: number analyzed (Participants) | 92 | 92 | 184
    Infants: Hispanic or Latino | 3 | 7 | 10
    Infants: Not Hispanic or Latino | 88 | 85 | 173
    Infants: Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Race for some mothers and infants was not reported
  Participants
    Mothers: number analyzed (Participants) | 92 | 92 | 184
    Mothers: American Indian or Alaska Native | 0 | 0 | 0
    Mothers: Asian | 1 | 0 | 1
    Mothers: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Mothers: Black or African American | 78 | 84 | 162
    Mothers: White | 4 | 1 | 5
    Mothers: More than one race | 4 | 4 | 8
    Mothers: Unknown or Not Reported | 5 | 3 | 8
    Infants: number analyzed (Participants) | 92 | 92 | 184
    Infants: American Indian or Alaska Native | 1 | 0 | 1
    Infants: Asian | 1 | 0 | 1
    Infants: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Infants: Black or African American | 75 | 84 | 159
    Infants: White | 3 | 1 | 4
    Infants: More than one race | 6 | 6 | 12
    Infants: Unknown or Not Reported | 6 | 1 | 7
Region of Enrollment [Number; unit: participants] — Region of Enrollment for Mother participants Population: Analysis includes mother participants only
  participants
    United States: number analyzed (Participants) | 92 | 92 | 184
    United States | 92 | 92 | 184
Region of Enrollment [Number; unit: participants] — Region of Enrollment for Infant participants Population: Analysis includes infant participants only
  participants
    United States: number analyzed (Participants) | 92 | 92 | 184
    United States | 92 | 92 | 184

OUTCOME MEASURES:

1. Primary Outcome: PHQ9
Description: Depression symptoms; Patient Health Questionnaire-9; values = 0-27; higher scores = worse outcome
Time Frame: Pre-intervention at Baseline (T1 data collected); [Intervention Period (8 months)]; Post-intervention (T2 data collected; 1 month post intervention)
Population: Discrepancy between Participant Flow and analyzed number is due to missing data for analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
score on a scale
  Pre-intervention: number analyzed (Participants) | 70 | 79
  Pre-intervention | 11.94 (6.35) | 10.31 (6.74)
  Post-intervention: number analyzed (Participants) | 70 | 79
  Post-intervention | 5.61 (5.60) | 5.33 (5.85)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p = 0.503, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

2. Primary Outcome: Landry Parent Child Interaction Rating Scales - Mother Positive Behavior
Description: Rating scale used for coding observed parent and child behavior during semi-structured free play. Reported outcomes include:
  mother positive behavior (values = 4-20; higher scores = better outcomes);
Time Frame: as for outcome 1
Population: Numbers analyzed differ due to missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
score on a scale
  Pre-Intervention: number analyzed (Participants) | 63 | 73
  Pre-Intervention | 12.43 (3.72) | 13.16 (4.02)
  Post-Intervention: number analyzed (Participants) | 63 | 73
  Post-Intervention | 15.54 (3.10) | 13.04 (3.94)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p < 0.001, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

3. Primary Outcome: Landry Parent Child Interaction Rating Scales - Mother Negative Behavior
Description: Dichotomized rating scale used for coding observed parent and child behavior during semi-structured free play. Reported outcomes include:
  mother negative behavior (values = 0-1; higher scores = worse outcomes)
Time Frame: as for outcome 1
Population: Numbers analyzed differ due to missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
score on a scale
  Pre-Intervention: number analyzed (Participants) | 63 | 73
  Pre-Intervention | 0.27 (0.06) | 0.25 (0.05)
  Post-Intervention: number analyzed (Participants) | 63 | 73
  Post-Intervention | 0.21 (0.06) | 0.38 (0.05)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p = 0.059, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

4. Primary Outcome: Landry Parent Child Interaction Rating Scales - Child Positive/Engagement Behavior
Description: Rating scale used for coding observed parent and child behavior during semi-structured free play. Reported outcomes include:
  child positive/engagement behavior (values = 2-10; higher scores = better outcomes)
Time Frame: as for outcome 1
Population: Numbers analyzed differ due to missing data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
score on a scale
  Pre-Intervention: number analyzed (Participants) | 63 | 73
  Pre-Intervention | 5.21 (1.94) | 4.97 (1.99)
  Post-Intervention: number analyzed (Participants) | 63 | 73
  Post-Intervention | 6.35 (2.20) | 5.92 (1.95)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p = 0.702, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

5. Primary Outcome: Indicator of Parent Child Interaction (IPCI) - Mother Maintain/Extend
Description: Direct observation, semi-structured direct infant-mother interaction looking at books. Reported includes:
  Mother Maintain/Extend (values = 0-100%; higher = better outcomes);
Time Frame: as for outcome 1
Population: Number analyzed differs due to missing data
Measure: Mean (Standard Deviation); unit: percentage of occurrence
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
percentage of occurrence
  Pre-intervention: number analyzed (Participants) | 60 | 71
  Pre-intervention | 1.92 (6.0) | 3.45 (7.54)
  Post-intervention: number analyzed (Participants) | 60 | 71
  Post-intervention | 5.83 (13.02) | 3.66 (7.22)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p = 0.08, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

6. Primary Outcome: Indicator of Parent Child Interaction (IPCI) - Mother Overall Positive
Description: Direct observation, semi-structured direct infant-mother interaction looking at books. Reported includes:
  Mother Overall Positive (values = 0-100%; higher = better outcomes)
Time Frame: as for outcome 1
Population: Number analyzed differs due to missing data
Measure: Mean (Standard Deviation); unit: percentage of occurrence
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
percentage of occurrence
  Pre-intervention: number analyzed (Participants) | 60 | 71
  Pre-intervention | 29.79 (15.46) | 30.39 (18.63)
  Post-intervention: number analyzed (Participants) | 60 | 71
  Post-intervention | 39.47 (18.54) | 33.54 (15.45)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p = 0.09, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

7. Primary Outcome: Indicator of Parent Child Interaction (IPCI) - Child Positive Social
Description: Direct observation, semi-structured direct infant-mother interaction looking at books. Reported includes:
  Child Positive Social (values = 0-100%; higher = better outcomes);
Time Frame: as for outcome 1
Population: Number analyzed differs due to missing data
Measure: Mean (Standard Deviation); unit: percentage of occurrence
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
percentage of occurrence
  Pre-intervention: number analyzed (Participants) | 60 | 71
  Pre-intervention | 16.50 (14.83) | 14.82 (14.29)
  Post-intervention: number analyzed (Participants) | 60 | 71
  Post-intervention | 27.96 (14.83) | 25.81 (18.16)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p = 0.898, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

8. Primary Outcome: Indicator of Parent Child Interaction (IPCI) - Child Engagement
Description: Direct observation, semi-structured direct infant-mother interaction looking at books. Reported includes:
  Child Engagement (values = 0-100%; higher = better outcomes)
Time Frame: as for outcome 1
Population: Number analyzed differs due to missing data
Measure: Mean (Standard Deviation); unit: percentage of occurrence
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
percentage of occurrence
  Pre-intervention | 31.14 (15.89) | 32.70 (14.40)
  Post-intervention | 42.44 (15.09) | 40.56 (16.78)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p = 0.349, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

9. Primary Outcome: Knowledge of Infant Social-Emotional Development and Promotion
Description: Rating scale used to assess understanding of the concepts of infant social-emotional behavior and its promotion by caregivers, assessing both definitional and applied concept knowledge; values = 0-28 higher scores = better outcomes
Time Frame: as for outcome 1
Population: Discrepancy between Participant Flow and analyzed number is due to missing data for analysis
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Mom & Baby Net | Depression & Developmental Awareness System
Number analyzed (Participants) | 92 | 92
score on a scale
  Pre-intervention: number analyzed (Participants) | 70 | 79
  Pre-intervention | 8.62 (0.45) | 8.01 (0.41)
  Post-intervention: number analyzed (Participants) | 70 | 79
  Post-intervention | 14.66 (0.56) | 8.54 (0.51)
Statistical Analysis 1: Comparison: Mom & Baby Net vs Depression & Developmental Awareness System; Test type: Superiority; p < 0.001, GLM Repeated Measures — P-value is Bonferroni correction adjusted at 0.05

ADVERSE EVENTS:
Time Frame: Pre-intervention at Baseline (T1 data collected); [Intervention Period (8 months)]; Post-intervention (T2 data collected; 1 month post intervention)
Groups:
- Mom & Baby Net Mothers; Mom & Baby Net Infants: CBT skills based mobile intervention targeting maternal depression and sensitive responsive parenting practices for optimizing infant social-communication promotion and provision of community resources and referral
  Mom & Baby Net: CBT skills based mobile intervention targeting maternal depression and sensitive responsive parenting practices for optimizing infant social-communication promotion and provision of community resources and referral
- Depression & Developmental Awareness System Mothers; Depression & Developmental Awareness System Infants: Supportive, person-centered mobile intervention targeting maternal awareness of maternal depression symptoms, infant developmental milestones, and provision of community resources and referral (active control condition)
  Depression & Developmental Awareness System: Supportive, person-centered mobile intervention targeting maternal awareness of maternal depression symptoms, infant developmental milestones, and provision of community resources and referral (active control condition)
Arm/Group | Mom & Baby Net Mothers | Depression & Developmental Awareness System Mothers | Mom & Baby Net Infants | Depression & Developmental Awareness System Infants
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92 | 0/92 | 0/92
Serious Adverse Events (participants affected / at risk) | 0/92 | 0/92 | 0/92 | 0/92
Other Adverse Events (participants affected / at risk) | 0/92 | 0/92 | 0/92 | 0/92

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Informed Consent Form (2018-11-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT03464630/Prot_ICF_002.pdf
  • Statistical Analysis Plan (2016-09-18): https://cdn.clinicaltrials.gov/large-docs/30/NCT03464630/SAP_001.pdf